CLINICAL TRIAL: NCT03613558
Title: A Double Blinded Randomized Placebo Controlled Study Evaluating the Use of Intraoperative Dexmedetomidine in Reducing Postoperative Pain and Narcotic Requirement in Patients With Moderate to Severe OSA.
Brief Title: Dex as Analgesic Adjuvant in OSA Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to recruit patients because the surgeon left the hospital
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-10-168
Record Dates: First submitted 2018-03-20; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Dexmedetomidine
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- Dexmedetomidine Sedation (Experimental): This group will receive 1mcg/kg bolus of dexmedetomidine over 15 minutes after intubation followed by an infusion of dexmedetomidine at 0.5mcg/kg/hr until approximately 30 minutes before the end of surgery.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): This group will receive a colorless, odorless liquid (i.e. normal saline) in order to resemble Dexmedetomidine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is an alpha-2 agonist that provides both sedation and analgesia
  Other Names: Precedex
  Arms: Dexmedetomidine Sedation
Drug: Placebo — saline solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether intravenous peri-operative Dexmedetomidine reduces opioid requirements and or improves pain control after Uvulopalatopharyngoplasty (UPPP) in patients with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
BACKGROUND/STUDY SIGNIFICANCE

Patients with OSA undergoing surgery have increased surgical risk compared to patients that do not have OSA . Perioperative medication such as benzodiazepines and opioids can decrease upper airway tone, inhibit central respiratory drive and inhibit upper airway reflexes. The supine position may also worsen the severity of the OSA. Additionally, this group of patients is more likely to have a higher incidence of complications, particularly post operative hypoxemia , difficult intubation , and complicated extubation course .

Uvulopalatopharyngoplasty (UPPP) along with other tongue base procedures are commonly performed surgical procedures used to help alleviate the symptoms of obstructive sleep apnea (OSA). Postoperative management of oropharyngeal pain is challenging since narcotic administration may compromise respiratory status in OSA patients. The Anesthesiology and Otorhinolaryngology communities have begun to rethink acceptable narcotic use in OSA patients especially following the recent FDA announcement highlighting serious adverse effects related to codeine consumption in children who had undergone tonsillectomies.

Dexmedetomidine (Precedex) is a sedative with minimal respiratory depression. Its mechanism is via alpha 2 agonism and has 8 times the affinity for the alpha 2 adrenoreceptor than clonidine. It has been shown to have sedative, analgesic, and anxiolytic effects. It produces a predictable and dose dependent decrease in heart rate and blood pressure. Dexmedetomidine undergoes extensive metabolism in the liver and is then eliminated as methyl and glucuronide conjugates mostly via the renal system. The pharmacokinetics are markedly affected by hepatic insufficiency .

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients scheduled for UPPP
* Patients with diagnosis of OSA via polysomnography
* American Society of Anesthesiology (ASA) classification 3 or lower

Exclusion Criteria:

* Bradycardia as defined as resting heart rate <60 Beats per min (BPM) or symptomatic
* Any degree of heart block diagnosed by ECG
* Hypotension as defined as <20% from baseline or symptomatic
* Liver failure, (two fold rise in liver enzymes)
* Chronic Kidney Disease (CKD) III or greater
* History of allergy to opioids or dexmedetomidine
* ASA classification 4 or higher
* ICU or Step down admission
* Difficult airway as defined by previous history of difficult intubation or requiring a fiberoptic intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Pain Score | within 24 hours post-operative
  Patient self-reported pain scores will be measured immediately after awakening post-op using the Numerical Pain Rating Scale and opioid requirements using morphine equivalents

SECONDARY OUTCOMES:
Pain Score | within 24 hours post-operative
  Pain score and opioid requirements will continue to be measured up to 24 hours postoperatively
Nausea | within 24 hours post-operative
  participants experience of nausea will be reported
Hypoxia | within 24 hours post-operative
  Number of hypoxic events will be calculated
Length of hospital stay | from admission to discharge, up to 14 days
  Number of days spent in the hospital from admission to discharge will be assessed.
Sedation | within 24 hours post-operative
  Ramsay Sedation Scale
Time to extubation | from post-operative until extubation, up to 72 hours
  length of time from operation to removal of endotracheal tube will be measured
Number of participants experiencing vomiting | within 24 hours post-operative
  participants' experiencing vomiting will be assessed and reported by care providers

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Straker, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Young T, Palta M, Dempsey J, Peppard PE, Nieto FJ, Hla KM. Burden of sleep apnea: rationale, design, and major findings of the Wisconsin Sleep Cohort study. WMJ. 2009 Aug;108(5):246-9. PMID 19743755
- [Background] Hillman DR, Loadsman JA, Platt PR, Eastwood PR. Obstructive sleep apnoea and anaesthesia. Sleep Med Rev. 2004 Dec;8(6):459-71. doi: 10.1016/j.smrv.2004.07.002. PMID 15556378
- [Background] Kaw R, Pasupuleti V, Walker E, Ramaswamy A, Foldvary-Schafer N. Postoperative complications in patients with obstructive sleep apnea. Chest. 2012 Feb;141(2):436-441. doi: 10.1378/chest.11-0283. Epub 2011 Aug 25. PMID 21868464
- [Background] Siyam MA, Benhamou D. Difficult endotracheal intubation in patients with sleep apnea syndrome. Anesth Analg. 2002 Oct;95(4):1098-102, table of contents. doi: 10.1097/00000539-200210000-00058. PMID 12351303
- [Background] Reeder MK, Goldman MD, Loh L, Muir AD, Casey KR, Gitlin DA. Postoperative obstructive sleep apnoea. Haemodynamic effects of treatment with nasal CPAP. Anaesthesia. 1991 Oct;46(10):849-53. doi: 10.1111/j.1365-2044.1991.tb09599.x. PMID 1952000
- [Background] Bhana N, Goa KL, McClellan KJ. Dexmedetomidine. Drugs. 2000 Feb;59(2):263-8; discussion 269-70. doi: 10.2165/00003495-200059020-00012. PMID 10730549
- [Background] Farag E, Ghobrial M, Sessler DI, Dalton JE, Liu J, Lee JH, Zaky S, Benzel E, Bingaman W, Kurz A. Effect of perioperative intravenous lidocaine administration on pain, opioid consumption, and quality of life after complex spine surgery. Anesthesiology. 2013 Oct;119(4):932-40. doi: 10.1097/ALN.0b013e318297d4a5. PMID 23681143
- [Background] Berger R, Hsu JC. Bioequivalence trials, intersection-union tests and equivalence confidence sets. Statis Sci. 1996;11:283-319
- [Background] American Academy of Sleep Medicine. International classification of sleep disorders, 2nd ed: Diagnostic and coding manual, American Academy of Sleep Medicine, Westchester, IL 2005.
- [Background] FDA. (2012, August 15) FDA Drug Safety Communication: Codeine use in certain children after tonsillectomy and/or adenoidectomy may lead to rare, but life-threatening adverse events or death. FDA.gov Retrieved August 8, 2013 from http://www.fda.gov/Drugs/DrugSafety/ucm313631.htm#safety.